CLINICAL TRIAL: NCT04851093
Title: Effects of Traditional Chinese Medicine on AECOPD Risk Window Patients: A Multi-center, Randomized, Double-blind, Controlled Trial
Brief Title: Effects of Traditional Chinese Medicine on Outcomes in Patients With AECOPD Risk Window
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCM for AECOPD Risk Window
Record Dates: First submitted 2021-04-01; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Acute Exacerbation Risk Window; Traditional Chinese Medicine; Randomized Controlled Trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM granule plus conventional drug (Experimental): The experimental group will receive three types of TCM granule and conventional drug according to 2020 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and Chinese Medicine Diagnosis Treatment Guidelines.
  Interventions: Drug: TCM granule plus conventional drug
- TCM placebo granule plus conventional drug (Placebo Comparator): The control group will receive three types of TCM placebo granule and conventional drug according to 2020 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and Chinese Medicine Diagnosis Treatment Guidelines.
  Interventions: Drug: TCM placebo granule plus conventional drug

INTERVENTIONS:
Drug: TCM granule plus conventional drug — All patients will receive conventional drug according to 2020 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and Chinese Medicine Diagnosis Treatment Guidelines.
  Yiqiwenfei granule for qi deficiency and internal cold fluid syndrome.
  Fuzhengqinghua granule for qi and yin deficiency and unclean phlegm heat syndrome.
  Fuzhengzaohua granule for lung and spleen qi deficiency and phlegm-damp amassing in lung syndrome.
  TCM granule (Jiangyin Tian Jiang Pharmaceutical Co.,Ltd, 10g/packet) will be administered twice daily for 8 weeks.
  Arms: TCM granule plus conventional drug
Drug: TCM placebo granule plus conventional drug — All patients will receive conventional drug according to 2020 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and Chinese Medicine Diagnosis Treatment Guidelines.
  Placebo Yiqiwenfei granule for qi deficiency and internal cold fluid syndrome.
  Placebo Fuzhengqinghua granule for qi and yin deficiency and unclean phlegm heat syndrome.
  Placebo Fuzhengzaohua granule for lung and spleen qi deficiency and phlegm-damp amassing in lung syndrome.
  TCM placebo granule (Jiangyin Tian Jiang Pharmaceutical Co.,Ltd, 10g/packet) will be administered twice daily for 8 weeks.
  The appearance, weight, color and odor of the preparation are the same as those of experimental group.
  The placebo granule consists of dextrin, bitter and 5% of the TCM granule.
  Arms: TCM placebo granule plus conventional drug

SUMMARY:
This study aims to objectively evaluate the clinical efficacy and safety of Traditional Chinese Medicine in the treatment of AECOPD Risk Window, providing a basis for the formulation of TCM treatment plan with AECOPD.

DETAILED DESCRIPTION:
The incidence, mortality, and prevalence of chronic obstructive pulmonary disease (COPD) are high, with a prevalence among people 40 years of age or older of 10.1% worldwide and 13.7% in China. COPD has become the third leading cause of death worldwide. Acute exacerbations of COPD (AECOPD) are important events in the management of COPD because they negatively impact health status, readmission, and disease progression.

Due to the non-random and non-accidental occurrence of AECOPD，with acute exacerbations occurring mainly in a centralized period after an acute exacerbation, and wide open to attack easily in this period, we call this "highly dangerous period" as "AECOPD Risk Window". The AECOPD Risk Window has persistent systemic inflammation and unstable lung function, which increases the risk of AECOPD recurrence and readmission.

At present, western medicine has relatively mature treatment measures for COPD at the acute exacerbation stage and stable stage, however, there is no specific guidance on the medication of AECOPD Risk Window. COPD have been effectively treated with Chinese medicine for a long time. The study of syndrome regularity of "AECOPD Risk Window" provides a basis for the formulation of syndrome differentiation plan.

This is a multi-center, randomized, double-blind, controlled trial to compare the efficacy of two therapies for patients with AECOPD Risk Window. 336 subjects will be randomly assigned in a 1:1 ratio to experimental group or control group for 8 weeks treatment and 18 weeks follow-up. On the basis of health education and conventional treatment, the experimental group will receive TCM granule according to the TCM syndrome, while the control group will receive TCM placebo granule according to the TCM syndrom. The primary outcomes are acute exacerbation rate in the AECOPD Risk Window, COPD Assessment Test (CAT) in the AECOPD Risk Window; and secondary outcomes are time to the first acute exacerbation, degree of acute exacerbation in the AECOPD Risk Window, acute exacerbation rate in the follow-up period, degree of acute exacerbation in the follow-up period, COPD Assessment Test (CAT) in the follow-up period, lung function, clinical symptom scores, mMRC, quality of life and index of security.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of AECOPD Risk Window;
2. Age ranges from 40 years to 80 years;
3. Syndrome differentiation meets criteria of qi deficiency and internal cold fluid syndrome, qi and yin deficiency and unclean phlegm heat syndrome, or lung and spleen qi deficiency and phlegm-damp amassing in lung syndrome;
4. Without participations in other interventional trials in the previous one month;
5. With the informed consent signed.

Exclusion Criteria:

1. Pregnant and lactating women;
2. Dementia, mental disorders and reluctant partners;
3. Complicated with heart failure (NYHA Class IV), or Serious cardiac arrhythmias, or unstable hemodynamics;
4. Current respiratory disorders other than COPD (e.g., bronchiectasis, active tuberculosis, pneumothorax, Pleural effusion, pulmonary thromboembolic, or Neuromuscular diseases affect respiratory movement function);
5. Complicated with serious hepatic and renal diseases (liver cirrhosis, portal hypertension, bleeding of varicose veins, dialysis, or renal transplantation);
6. Bedridden for various reasons;
7. Allergic to the used medicine.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute exacerbation rate in the AECOPD Risk Window | in 8 weeks of the treatment period.
  The numbers of acute exacerbation in the AECOPD Risk Window will be recorded.
COPD Assessment Test (CAT) in the AECOPD Risk Window | Change from baseline CAT scores at week 0, 8 of the treatment period.
  The COPD assessment test (CAT) is a self-administered questionnaire that measures health-related quality of life. It is an 8-item questionnaire on a 0-5 point scale with higher values indicating greater impact of COPD. The item response values of CAT are summed to produce a single score that ranges from 0-9 (low impact), 10-20 (medium impact), 21-30 (high impact) and 31-40 (very high impact).

SECONDARY OUTCOMES:
Time to the first acute exacerbation | up to week 26 during the study period.
  Time from the first exacerbation to the last exacerbation will be recorded.
Degree of acute exacerbation in the AECOPD Risk Window | in 8 weeks of the treatment period.
  The numbers of acute exacerbation of different severity in the AECOPD Risk Window will be recorded..
Acute exacerbation rate in the follow-up period | in 18 weeks of the follow-up period.
  The numbers of acute exacerbation in the follow-up period will be recorded.
Degree of acute exacerbation in the follow-up period | in 18 weeks of the follow-up period.
  The numbers of acute exacerbation of different severity in the follow-up period will be recorded.
COPD Assessment Test (CAT) in the follow-up period | Change from baseline CAT scores at week 16, 26 of the follow-up period.
  The COPD assessment test (CAT) is a self-administered questionnaire that measures health-related quality of life. It is an 8-item questionnaire on a 0-5 point scale with higher values indicating greater impact of COPD. The item response values of CAT are summed to produce a single score that ranges from 0-9 (low impact), 10-20 (medium impact), 21-30 (high impact) and 31-40 (very high impact).
Pulmonary function | at week 0, 8 of the treatment period and at week 26 of the follow-up period.
  The Forced expiratory volume in one second ( FEV1), Forced Vital Capacity (FVC), FEV1% (FEV1/FVC) will be used to assess pulmonary function.
Clinical symptom scores | Change from baseline clinical symptom scores at week 0, 8 of the treatment period and at week 16, 26 of the follow-up period.
  Clinical symptom scores of COPD will be used to assess symptoms. The clinical symptoms to be evaluated in this study include cough, expectoration, wheezing, chest tightness, shortness of breath, and fatigue. A score of 0-3 will be given to every symptom or sign with a higher score indicating a worse conditoin.
mMRC | Change from baseline mMRC scores at week 0, 8 of the treatment period and at week 16, 26 of the follow-up period.
  The modified Medical Research Council (mMRC) scale is a 5-point (0-4) scale based on the severity of dyspnoea. "0" means no dyspnea perception, "4" means severe dyspnea perception.
SGRQ | Change from baseline SGRQ scores at week 0, 8 of the treatment period and at week 16, 26 of the follow-up period.
  The St. George's Respiratory Questionnaire (SGRQ) scores will be used to evaluate quality of life with a total score of 0-100. The higher scores will indicate the worse outcomes.
mCOPD-PRO | Change from baseline mPRO-COPD scores at week 0, 8 of the treatment period and at week 16, 26 of the follow-up period
  The modified COPD Patient-Reported Outcome scale (mCOPD-PRO) will be used to assess quality of life. The mCOPD-PRO contains 27 items in three domains. mCOPD-PRO scores range from 0 to 4 with a decrease in score showing higher health status.
mESQ-COPD | Change from baseline mESQ-COPD scores at week 0, 8 of the treatment period and at week 16, 26 of the follow-up period.
  The modified Effectiveness Satisfaction Questionnaire for COPD (mESQ-COPD) will be used to assess treatment satisfaction. The mESQ-COPD contains 19 items in four domains. mESQ-COPD scores range from 0 to 4 with a decrease in score showing higher treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, doctor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China